CLINICAL TRIAL: NCT03530176
Title: 18F-Sodium Fluoride (18F-NaF) PET-CT Imaging to Identify Vulnerable Plaques in Patients With Diabetes
Acronym: D-NaF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Paolo Raggi, MD, Section Chief of Cardiology, Mazankowski Alberta Heart Institute, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00049579
Record Dates: First submitted 2016-09-16; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Atherosclerosis; Complications of Diabetes Mellitus
MeSH Terms: conditions — Atherosclerosis; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): 18F-NaF (sodium Flouride ) is a radio-pharmaceutical used to image skeletal pathology, including primary and secondary neoplasms. Despite US Federal Drug Administration (FDA) approval and 18F-NaF being listed in the US Pharmacopeia, 18F-NaF is not currently approved by Health Canada for use as a cardiac imaging tracer. Therefore, a concurrent Health Canada Clinical Trial Application is being submitted to ensure its availability. Intervention on single arm: A dose of 18F-NaF (200 - 400 MBq) will be injected intravenously at rest. After a 60 minute, an ECG-gated PET acquisition will be performed centered over the heart for 20 minutes. A CT coronary calcium score examination will also be performed on a dedicated CT scanner and the Agatston and volume scores calculated according to standards.
  Interventions: Radiation: 18Fluoride-Sodium Fluoride radio-isotope

INTERVENTIONS:
Radiation: 18Fluoride-Sodium Fluoride radio-isotope — The investigators will be using 18F-NaF to image premature atherosclerosis in the coronary arteries of diabetic patients.
  Other Names: 18F-NaF

SUMMARY:
Coronary artery calcification is a sign of heart disease. A nuclear medicine PET-CT test using sodium fluoride (18F-NaF) radioisotope has been shown to help identify growing calcification plaques early on in the disease process. It is known that diabetic patients are at a high risk of developing premature coronary disease; the investigators intend to use this new technology to identify those patients at higher risk of developing coronary artery disease.

DETAILED DESCRIPTION:
Diabetic patients are at very high risk of suffering premature coronary artery disease events compared to the general population. Whether pancreas transplant completely reverses the biochemical imbalances of diabetes mellitus and the high cardiovascular risk of these patients is unclear. Investigators in the field of imaging have been looking for ways to identify patients at greater risk of suffering events by searching for plaques in the cardiovascular system more likely to fracture and cause acute intravascular thrombosis (vulnerable plaques) with subsequent precipitation of acute events. Recent advances in PET-CT provide an opportunity to pursue such search with limited risk to the patient and high probability of success. CT scanning is used to identify vascular calcification -a marker of atherosclerosis- and PET imaging with 18F-NaF helps determine whether the calcification is actively accumulating calcium and phosphorus making it an actively growing plaque. PET imaging with 18F-NaF has been used in the setting of acute coronary syndromes to identify the most active and unstable plaques and in patients with severe aortic valve stenosis to follow the natural history of this disease. The investigators propose to perform PET-CT imaging with 18F-NaF in a pilot study of 100 patients chosen among the subjects followed in the outpatient diabetes clinics at the University of Alberta. The aim is to investigate the presence and extent of unstable plaques in ambulatory patients affected by diabetes, and to identify a set of clinical variables most likely to be associated with a large burden of disease. Since there are no published studies in this particular field it is impossible to make precise sample size calculations and these analyses must therefore be considered exploratory.

ELIGIBILITY:
Inclusion Criteria:

> 18 years of age. Has an established diagnosis of diabetes mellitus type 1 or 2. Stable clinical course with a stable medical regimen for 6 months prior to enrollment.

-

Exclusion Criteria:

Unable to give consent. Weight >250 kg. Unable to lie flat for 20-30 minutes to complete the PET-CT session. Pregnancy, breast feeding, known history of primary hyperparathyroidism or metabolic bone disease, recent malignancy (<3 years) or previous thoracic irradiation.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
18F-Sodium Fluoride (18F-NaF) PET-CT Imaging to Identify Vulnerable Plaques in Patients With Diabetes | 4-6 weeks
  Prevalence of patients with type-2 diabetes and unstable, high-risk coronary artery plaques

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Raggi, MD, Principal Investigator — Professor of Medicine, University of Alberta
Locations (1):
- University Hospital of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raggi P, Senior P, Shahbaz S, Kaul P, Hung R, Coulden R, Yeung R, Abele J. 18F-Sodium Fluoride Imaging of Coronary Atherosclerosis in Ambulatory Patients With Diabetes Mellitus. Arterioscler Thromb Vasc Biol. 2019 Feb;39(2):276-284. doi: 10.1161/ATVBAHA.118.311711. PMID 30580559